CLINICAL TRIAL: NCT01316055
Title: A Parallel, Three Arm, Open-label, Multi-dose Pharmacokinetic Study of Dalfampridine-ER 7.5 mg Twice Daily in Both Healthy Volunteers and Those With Mild and Moderate Renal Impairment
Brief Title: Pharmacokinetics (PK) of Dalfampridine-ER 7.5 mg BID in Healthy Volunteers and Subjects With Mild or Moderate Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RD7.5D-ER012010
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Results first posted 2012-11-07 (Estimated); Last update posted 2012-11-07 (Estimated); Status verified 2012-10

CONDITIONS: Renal Insufficiency
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy: Dalfampridine-ER 7.5 mg (Active Comparator): Dalfampridine-ER 7.5 mg single and steady-state dosing in healthy volunteers
  Interventions: Drug: Dalfampridine-ER
- Mild renal: Dalfampridine-ER 7.5 mg (Active Comparator): Dalfampridine-ER 7.5 mg single and steady-state dosing in volunteers with mild renal impairment
  Interventions: Drug: Dalfampridine-ER
- Moderate renal: Dalfampridine-ER 7.5 mg (Active Comparator): Dalfampridine-ER 7.5 mg single and steady-state dosing in volunteers with moderate renal impairment
  Interventions: Drug: Dalfampridine-ER

INTERVENTIONS:
Drug: Dalfampridine-ER — 2 days of single dose 7.5 mg, 4 days of bid dosing, and a 3 day follow-up

SUMMARY:
The steady-state pharmacokinetics of Dalfampridine-ER (extended release) 7.5 mg (milligram) tablets in healthy adult volunteers and those with mild and moderate renal impairment, and examine between group comparisons.

DETAILED DESCRIPTION:
Pharmacokinetics in normal, mildly renally impaired, and moderately renally impaired subjects

ELIGIBILITY:
Inclusion Criteria:

* Either gender between the ages of 18 and 75 years
* Have a body mass index (BMI) ranging between 18.5 - 35.0 kg/m2, inclusive
* Have adequate cognitive function to understand and sign the IRB approved informed consent prior to the performance of any study-specific procedures
* Be willing and able to comply with all trial requirements
* Fit into one of three 12-subject groups: normal renal function (CrCl > 80 mL/min), mild renal impairment (CrCl 51-80 mL/min), and moderate renal impairment (CrCl 30-50 mL/min)
* Have sufficient venous access to permit blood sample collection
* Women of childbearing potential must have a negative β-HCG pregnancy test at the Screening Visit.

Exclusion Criteria:

* Women who are either pregnant or breastfeeding, and women of childbearing potential (i.e., has not had a hysterectomy or bilateral oophorectomy, or is not at least two years postmenopausal) who are engaged in active heterosexual relations and not using any of the following birth control methods: tubal ligation, implantable contraception device, oral, patch or injectible contraceptive, double barrier method, or sexual activity restricted to a vasectomized partner;
* History of seizure(s);
* Unstable, acute, or severe (CrCl < 30 mL/min) renal failure;
* Clinically significant abnormal findings on the physical examination, ECG, vital signs, medical history, or clinical laboratory results during screening (other than abnormal renal values);
* Any unstable cardiovascular, enterohepatic, respiratory, or immunologic disorder or disease that may substantially affect the pharmacokinetics of Dalfampridine-ER;
* Known allergy to pyridine-containing substances, or any of the inactive ingredients of the Dalfampridine-ER tablet (colloidal silicon dioxide, hydroxypropyl methylcellulose, magnesium stearate, microcrystalline cellulose, polyethylene glycol, and titanium dioxide);
* Participation in an investigational drug trial 30 days prior to Screening or plans to enroll in an investigational drug trial at any time during this study;
* Any medical condition including psychiatric disease that would interfere with the interpretation of the study results or the conduct of the study;
* Subject has started a new medication (prescription, vitamins, herbal medications, or other over-the-counter medications), or had a change in their existing medication within 30 days prior to screening;
* History of drug or alcohol abuse in the past 2 years, or tests positive for drugs of abuse at Screening;
* Donation of blood or blood components within 30 days prior to administration of investigational drug. The Investigator should instruct subjects who participate in this study not to donate blood or blood components during their participation in the study and up to four weeks after the completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-01; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert R Henney, PharmD, Study Director — Acorda Therapeutics
Locations (2):
- United States (2):
  - ACRI - Phase 1, Anaheim, California
  - MRA Clinical Research, South Miami, Florida

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject screened January, 2011. Last subject out August, 2011. Full Service Phase 1 Units.
Groups:
- Healthy: Dalfampridine-ER 7.5 mg: Dalfampridine-ER 7.5 mg single and steady-state dosing in healthy volunteers
  Dalfampridine-ER : 2 days of single dose 7.5 mg, 4 days of bid dosing, and a 3 day follow-up
- Mild Renal: Dalfampridine-ER 7.5 mg: Dalfampridine-ER 7.5 mg single and steady-state dosing in volunteers with mild renal impairment
  Dalfampridine-ER : 2 days of single dose 7.5 mg, 4 days of bid dosing, and a 3 day follow-up
- Moderate Renal: Dalfampridine-ER 7.5 mg: Dalfampridine-ER 7.5 mg single and steady-state dosing in volunteers with moderate renal impairment
  Dalfampridine-ER : 2 days of single dose 7.5 mg, 4 days of bid dosing, and a 3 day follow-up
Period: Overall Study
Arm/Group | Healthy: Dalfampridine-ER 7.5 mg | Mild Renal: Dalfampridine-ER 7.5 mg | Moderate Renal: Dalfampridine-ER 7.5 mg
Started | 13 | 17 | 12
Completed | 12 | 17 | 12
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy: Dalfampridine-ER 7.5 mg | Mild Renal: Dalfampridine-ER 7.5 mg | Moderate Renal: Dalfampridine-ER 7.5 mg | Total
Number analyzed (Participants) | 13 | 17 | 12 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 2 | 23
  >=65 years | 2 | 7 | 10 | 19
Age Continuous [Mean (Standard Deviation); unit: years] | 41.9 (14.65) | 63.2 (7.22) | 67.1 (7.65) | 57.7 (14.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 7 | 4 | 14
  Male | 10 | 10 | 8 | 28
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 4 | 2 | 6
  Black or African American | 1 | 2 | 2 | 5
  White | 11 | 11 | 8 | 30
  Other | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Steady State Area Under the Drug Concentration Time Curve From 0 to 12 Hours Post Dose AUC(0-12).
Description: AUC(0-12) was based on blood samples taken at specified outcome measure time frame for dalfampridine-ER 7.5 mg tablets in healthy adult volunteers and people with mild or moderate renal impairment.
Time Frame: 0 and 1,2,3,4,5,6,8, and 12 hours after the last dose
Population: Intention to treat (ITT)
Measure: Geometric Mean (90% Confidence Interval); unit: hour*nanogram/milliliter
Arm/Group | Healthy: Dalfampridine-ER 7.5 mg | Mild Renal: Dalfampridine-ER 7.5 mg | Moderate Renal: Dalfampridine-ER 7.5 mg
Number analyzed (Participants) | 12 | 17 | 12
hour*nanogram/milliliter | 157.8 [130.4 to 190.9] | 276.5 [241.5 to 316.7] | 415.3 [383.8 to 449.4]

2. Secondary Outcome: The Maximum Measured Plasma Concentration (Cmax) at Steady State, of Dalfampridine-ER 7.5 mg Tablets in Healthy Adult Volunteers and Those With Mild and Moderate Renal Impairment and Examine Between-group Differences.
Time Frame: 7 days
Population: ITT
Measure: Geometric Mean (90% Confidence Interval); unit: nanogram/milliliter
Arm/Group | Healthy: Dalfampridine-ER 7.5 mg | Mild Renal: Dalfampridine-ER 7.5 mg | Moderate Renal: Dalfampridine-ER 7.5 mg
Number analyzed (Participants) | 12 | 17 | 12
nanogram/milliliter | 20.61 [17.76 to 23.92] | 33.92 [29.92 to 38.47] | 46.69 [43.68 to 49.91]

3. Secondary Outcome: The Steady State Fractional Clearance, Calculated as the Dose / AUC(0-12) (CL/Fss) of Dalfampridine-ER 7.5 mg Tablets in Healthy Adult Volunteers and Those With Mild and Moderate Renal Impairment and Examine Between-group Differences.
Time Frame: 7 days
Population: ITT
Measure: Geometric Mean (90% Confidence Interval); unit: liter/hour
Groups:
- Healthy: Dalfampridine-ER 7.5 mg: Dalfampridine-ER 7.5 mg steady-state dosing in healthy volunteers
  Dalfampridine-ER : 2 days of single dose 7.5 mg, 4 days of bid dosing, and a 3 day follow-up
- Mild Renal: Dalfampridine-ER 7.5 mg: Dalfampridine-ER 7.5 mg and steady-state dosing in volunteers with mild renal impairment
  Dalfampridine-ER : 2 days of single dose 7.5 mg, 4 days of bid dosing, and a 3 day follow-up
- Moderate Renal: Dalfampridine-ER 7.5 mg: Dalfampridine-ER 7.5 mg steady-state dosing in volunteers with moderate renal impairment
  Dalfampridine-ER : 2 days of single dose 7.5 mg, 4 days of bid dosing, and a 3 day follow-up
Arm/Group | Healthy: Dalfampridine-ER 7.5 mg | Mild Renal: Dalfampridine-ER 7.5 mg | Moderate Renal: Dalfampridine-ER 7.5 mg
Number analyzed (Participants) | 12 | 17 | 12
liter/hour | 47.54 [39.29 to 57.52] | 27.12 [23.68 to 31.06] | 18.06 [16.69 to 19.54]

ADVERSE EVENTS:
Time Frame: Total study participation was to last for approximately 7 days consisting of 2 in-clinic confinement periods (exclusive of up to 14 days of screening), and follow-up 3 days post final discharge.
Description: All adverse events with an onset time after dosing and up to 72 hours after the last dose of study drug were considered treatment-emergent. In addition, adverse events with onset date before start of trial treatment but with worsening in intensity during the treatment period were also considered treatment-emergent.
Arm/Group | Healthy: Dalfampridine-ER 7.5 mg | Mild Renal: Dalfampridine-ER 7.5 mg | Moderate Renal: Dalfampridine-ER 7.5 mg
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/17 | 0/12
Other Adverse Events (participants affected / at risk) | 8/13 | 8/17 | 4/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Healthy: Dalfampridine-ER 7.5 mg (N=13) | Mild Renal: Dalfampridine-ER 7.5 mg (N=17) | Moderate Renal: Dalfampridine-ER 7.5 mg (N=12)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Any TEAEs (treatment emergent adverse effects) (General disorders) | 8 (10) | 8 (10) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.